CLINICAL TRIAL: NCT07007286
Title: A Real-World Study on Reducing the Risk of Liver Cancer in Chronic Hepatitis B Patients With a Family History of HBV-Related Liver Cancer.
Brief Title: Real-world Study on Liver Cancer Risk in Chronic Hepatitis B Patients With Family History of Liver Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Chief physician, Peking University First Hospital
Other Study IDs: 2025086
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: HBV; HCC
MeSH Terms: interventions — TMF protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect blood samples as needed for omics testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEG IFNα-2b Group
  Interventions: Drug: ETV,TDF,TAF,TMF combination with PEG IFNα-2b
- Nucleos(t)ide Monotherapy Group
  Interventions: Drug: ETV,TDF,TAF or TMF

INTERVENTIONS:
Drug: ETV,TDF,TAF,TMF combination with PEG IFNα-2b — The study will not involve any additional interventions, nor will it interfere with any related clinical decision-making.
  Groups: PEG IFNα-2b Group
Drug: ETV,TDF,TAF or TMF — The study will not involve any additional interventions, nor will it interfere with any related clinical decision-making.
  Groups: Nucleos(t)ide Monotherapy Group

SUMMARY:
This study is a prospective, multicenter, real-world cohort study designed to compare the long-term outcomes of chronic hepatitis B patients with a family history of HBV-related hepatocellular carcinoma (HCC) who receive PEG IFNα-2b combined with nucleos(t)ide analogues or nucleos(t)ide monotherapy. The primary endpoint is the incidence rate of HCC, and secondary endpoints include the rate of HBsAg seroclearance, changes in liver fibrosis, and survival rates. The study will last for 5 years and enroll approximately 15,000 patients, aiming to provide evidence-based optimization for CHB treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* (1) Chronic hepatitis B (CHB) patients with HBsAg positivity for over 6 months; (2) Family history of HBV-related hepatocellular carcinoma (HCC) (first- or second-degree relatives with HBV-related HCC); (3) Age ≥ 30 years, regardless of gender; (4) Based on real-world clinical practice, patients receiving nucleos(t)ide analogue (NA) therapy, such as Entecavir (ETV), Tenofovir Disoproxil Fumarate (TDF), Tenofovir Alafenamide Fumarate (TAF), or Tenofovir Amibufenamide (TMF), or those receiving combination therapy with nucleos(t)ide analogues and PEG IFNα-2b; (5) Negative pregnancy test within 24 hours before the first dose (for women of childbearing potential); (6) Voluntary participation, with the ability to understand and sign the informed consent form.

Exclusion Criteria:

* (1) Patients diagnosed with hepatocellular carcinoma (HCC) or malignancies in other organ systems prior to treatment; (2) Patients with contraindications to Peg IFN α-2b (refer to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2022 Edition) for details); (3) Patients in the immune-tolerant phase of HBV infection; (4) Patients scheduled for or with a history of organ transplantation; (5) Patients with hypersensitivity to interferon or any contraindication listed in the drug's prescribing information; (6) Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion criteria but do not meet the exclusion criteria were screened from multiple centers nationwide.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
5-year incidence of hepatocellular carcinoma (HCC) | From the start of antiviral treatment to 5 years of follow-up.

SECONDARY OUTCOMES:
HBsAg seroclearance rate | From the start of antiviral treatment to 5 years of follow-up.
HBeAg seroclearance rate | From the start of antiviral treatment to 5 years of follow-up.
HBV DNA level | From the start of antiviral treatment to 5 years of follow-up.
HBsAg level | From the start of antiviral treatment to 5 years of follow-up.
HBeAg level | From the start of antiviral treatment to 5 years of follow-up.
Proportion of patients with improved or progressed liver fibrosis | From the start of antiviral treatment to 5 years of follow-up.
Median time to cirrhosis | From the start of antiviral treatment to 5 years of follow-up.
Median time to decompensated cirrhosis | From the start of antiviral treatment to 5 years of follow-up.
Median time to HCC | From the start of antiviral treatment to 5 years of follow-up.
Overall survival (OS) | From the start of antiviral treatment to 5 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Ph.D, Principal Investigator — Peking University First Hospital
Locations (555):
- China (555):
  - Qitaihe Infectious Disease Hospital, Heilongjiang, Heilongjiang
  - Yizheng People's Hospital, Yizheng, Jiangsu
  - Changle County People's Hospital, Changle, Shandong
  - Juxian People's Hospital, Junxian, Shandong
  - Pingdu People's Hospital, Shandong, Pingdu, Shandong
  - Zouping People's Hospital, Zouping, Shandong
  - Huozhou Coal & Electricity Group General Hospital Co., Ltd., Huozhou, Shanxi
  - Huozhou People's Hospital, Huozhou Medical Group, Huozhou, Shanxi
  - Huozhou People's Hospital, Huozhou, Shanxi
  - Fenxi Mining Group Employees General Hospital, Jiexiu, Shanxi
  - Jiexiu Medical Group People's Hospital, Jiexiu, Shanxi
  - Anfu County People's Hospital, Anfu
  - Ankang Central Hospital, Ankang
  - Ankang Hospital of Traditional Chinese Medicine, Ankang
  - Anning Hospital of Traditional Chinese Medicine, Anning
  - Anqing First People's Hospital, Anqing
  - Anqing Municipal Hospital, Anqing
  - Anshan Infectious Disease Hospital, Anshan
  - Anyue County People's Hospital, Anyue
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Baise City
  - Baoding First Central Hospital, Baoding
  - Baoding People's Hospital, Baoding
  - Baotou Central Hospital, Baotou
  - China National Medicines (CNM) Northern Hospital, Baotou
  - The Third Staff Hospital of Baotou Steel Group, Baotou
  - Beihai People's Hospital, Beihai
  - Beijing Daxing District People's Hospital, Beijing
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Ditan Hospital, Beijing
  - Beijing Fangshan District First Hospital, Beijing
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing
  - Beijing Huaxin Hospital, Beijing
  - Beijing Liangxiang Hospital, Fangshan District, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Beijing You'an Hospital, Capital Medical University, Beijing
  - Beijing You'an Hospital, Beijing
  - Dongfang Hospital, Beijing University of Chinese Medicine, Beijing
  - Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Shunyi Hospital of Traditional Chinese Medicine, Beijing, Beijing
  - The Fifth Medical Center of PLA General Hospital, Beijing
  - Wangfu Hospital of Integrated Traditional Chinese and Western Medicine, Beijing
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Bengbu Fifth People's Hospital, Bengbu
  - Guzhen County Hospital of Traditional Chinese Medicine, Bengbu
  - Guzhen County People's Hospital, Bengbu
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - Benxi Sixth People's Hospital, Benxi
  - Beihai Tuberculosis Prevention and Treatment Hospital, Bihua
  - Binzhou Central Hospital, Binzhou
  - Binzhou People's Hospital, Binzhou
  - Bozhou Hospital of Traditional Chinese Medicine, Bozhou
  - Bozhou People's Hospital, Bozhou
  - Lixin County People's Hospital, Bozhou
  - Mengcheng First People's Hospital, Bozhou
  - Cangzhou Third Hospital, Cangzhou
  - The First Hospital of Jilin University, Changchun
  - Changji Branch of the First Affiliated Hospital of Xinjiang Medical University, Changji
  - Changji Hui Autonomous Prefecture People's Hospital, Changji
  - Changxing County People's Hospital, Changxing
  - Changzhi People's Hospital, Changzhi
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Changzhou Third People's Hospital, Changzhou
  - Yizheng People's Hospital, Changzhou
  - Chaoyang Fourth Hospital, Chaoyang
  - Kazuo County Central Hospital, Chaoyang
  - Chengdu Fifth People's Hospital, Chengdu
  - Chengdu Public Health Clinical Medical Center, Chengdu
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chifeng Baoshan Hospital, Chifeng
  - Chifeng Songshan Traditional Chinese Medicine & Mongolian Medicine Hospital, Chifeng
  - Chifeng Tumor Hospital, Chifeng
  - Chizhou People's Hospital, Chizhou
  - Mingguang People's Hospital, Chuzhou
  - Dali Bai Autonomous Prefecture People's Hospital, Dali
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Dandong Sixth People's Hospital, Dandong
  - Daqing Second Hospital, Daqing
  - China National Medicines & Health Products Datong Coal Mine Group General Hospital, Datong
  - Datong Fourth People's Hospital, Datong
  - Donggang Central Hospital, Donggang
  - Dongguan Eastern Central Hospital, Dongguan
  - Dongguan Ninth People's Hospital, Dongguan
  - Dongtai People's Hospital, Dongtai
  - Dongying Hospital of Traditional Chinese Medicine, Dongying
  - Dongying People's Hospital, Dongying
  - Shengli Oilfield Central Hospital, Dongying
  - Jianshi County People's Hospital, Enshi
  - Lichuan Traditional Chinese Medicine Hospital for Ethnic Minorities, Enshi
  - Ezhou Central Hospital, Ezhou
  - Fengcheng People's Hospital, Fengcheng
  - Fenyang Hospital, Fenyang
  - Foshan Hospital of Traditional Chinese Medicine, Foshan
  - Sanshui Hospital of Zhujiang Hospital, Southern Medical University, Foshan
  - Shunde Hospital Affiliated to Jinan University, Foshan
  - The Eighth Affiliated Hospital of Southern Medical University, Foshan
  - The Fourth People's Hospital of Foshan, Foshan
  - Fuxin Infectious Disease Hospital, Fuxin
  - Fuyang Fifth People's Hospital, Fuyang
  - Fuyang Hospital Affiliated to Anhui Medical University, Fuyang
  - Fuyang People's Hospital, Fuyang
  - Fuyang Second People's Hospital, Fuyang
  - Linquan County People's Hospital, Fuyang
  - Taihe County Hospital of Traditional Chinese Medicine, Fuyang
  - Jinxi County People's Hospital, Fuzhou
  - Lichuan County People's Hospital, Fuzhou
  - Linchuan District First People's Hospital, Fuzhou
  - Nanfeng County People's Hospital, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Dingnan County First People's Hospital, Ganzhou
  - Ganzhou Fifth People's Hospital, Ganzhou
  - Ganzhou People's Hospital, Ganzhou
  - Yudu County People's Hospital, Ganzhou
  - Gaomi People's Hospital, Gaomi
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Guangzhou Medical University Affiliated Panyu Central Hospital, Guangzhou
  - Huadu District People's Hospital, Guangzhou, Guangzhou
  - Nansha District People's Hospital, Guangzhou, Guangzhou
  - Panyu District Maternal and Child Health Hospital, Guangzhou, Guangzhou
  - Shijing People's Hospital, Baiyun District, Guangzhou, Guangzhou
  - The Fourth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou
  - Guilin Hospital of Traditional Chinese Medicine, Guilin
  - The Third People's Hospital of Guilin, Guilin
  - Xing'an County People's Hospital, Guilin
  - Hainan Provincial People's Hospital, Haikou
  - Hailin People's Hospital, Hailin
  - Hami Central Hospital, Hami
  - Xinjiang Production and Construction Corps 13th Division Hongxing Hospital, Hami
  - Handan Central Hospital, Handan
  - Handan First Hospital, Handan
  - Handan Fourth Hospital, Handan
  - Handan Infectious Disease Hospital, Handan
  - Linzhang County People's Hospital, Handan
  - Wei County People's Hospital, Handan
  - Yongnian District First People's Hospital, Handan
  - Hangzhou Xixi Hospital, Hangzhou
  - Lin'an District First People's Hospital, Hangzhou
  - Linping District Hospital of Traditional Chinese Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou
  - Chenggu County People's Hospital, Hanzhong
  - Hanbin District First Hospital, Hanzhong
  - Hanzhong Second People's Hospital, Hanzhong
  - Yang County People's Hospital, Hanzhong
  - Acheng District People's Hospital of Harbin, Harbin
  - Harbin First Hospital, Harbin
  - Harbin Sixth Hospital, Harbin
  - Heilongjiang Provincial Hospital, Harbin
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Gu'an County Hospital of Traditional Chinese Medicine, Hebei
  - Anhui Provincial Hospital, Hefei
  - Hefei First People's Hospital Binhu Branch, Hefei
  - Hefei First People's Hospital, Hefei
  - Hefei Second People's Hospital, Hefei
  - Hefei Third People's Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Hegang Infectious Disease Hospital, Hegang
  - Hegang Mining General Hospital, Hegang
  - Beian First People's Hospital, Heihe
  - Heihe First People's Hospital, Heihe
  - Hengshui Third People's Hospital, Hengshui
  - Hotan Prefecture Specialized Hospital for Infectious Diseases, Hetian
  - Heze Municipal Hospital, Heze
  - Hezhou People's Hospital, Hezhou
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Hohhot Second Hospital, Hohhot
  - Inner Mongolia Autonomous Region Hospital of Traditional Chinese Medicine, Hohhot
  - The 969th Hospital of the Joint Logistics Support Force, Hohhot
  - The Fourth Hospital of Inner Mongolia Autonomous Region, Hohhot
  - Hongze District People's Hospital, Huai'an
  - Huai'an Fifth People's Hospital, Huai'an
  - Huai'an Fourth People's Hospital, Huai'an
  - Huai'an No. 82 Hospital, Huai'an
  - Huainan First People's Hospital, Huainan
  - Huangshan Huangshan People's Hospital, Huangshan City
  - Huangshan People's Hospital, Huangshan City
  - Qimen County People's Hospital, Huangshan City
  - Xiuning County People's Hospital, Huangshan City
  - Daye People's Hospital, Huangshi
  - Huangshi Central Hospital, Huangshi
  - Huangshi Hospital of Traditional Chinese Medicine, Huangshi
  - Yangxin County People's Hospital, Huangshi
  - Huazhong University of Science and Technology, Hubei
  - Jiamusi Infectious Disease Hospital, Jiamusi
  - Jiangmen Central Hospital, Jiangmen
  - Xinhui People's Hospital, Jiangmen
  - Jianping County Hospital, Jianping
  - Tongji University Affiliated Oriental Hospital Jiaozhou, Jiaozhou
  - Affiliated Hospital of Beihua University, Jilin
  - Jilin City Infectious Disease Hospital, Jilin
  - Jilin Provincial Hepatobiliary Hospital, Jilin
  - Qingdao Jimo District People's Hospital, Jimo
  - Jinan People's Hospital, Jinan
  - Jiyang District Hospital of Traditional Chinese Medicine, Jinan
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan
  - Shandong Provincial Public Health Clinical Center, Jinan
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - The Second Hospital of Shandong University, Jinan
  - Gaoping People's Hospital, Jincheng
  - Jincheng People's Hospital, Jincheng
  - Jincheng Third People's Hospital, Jincheng
  - Zezhou County People's Hospital, Jincheng
  - Gong'an County People's Hospital, Jingzhou
  - Jingzhou Central Hospital, Jingzhou
  - The First People's Hospital of Jingzhou, Hubei, Jingzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - Jining Public Health Medical Center, Jining
  - Jinxiang County People's Hospital, Jining
  - Jinxian County People's Hospital, Jinxian
  - Jinzhong First People's Hospital, Jinzhong
  - Shanxi Coking Coal Fenxi Mining Group Employees General Hospital, Jinzhong
  - Jinzhou Central Hospital, Jinzhou
  - Jinzhou Infectious Disease Hospital, Jinzhou
  - Jiujiang Hospital of Traditional Chinese Medicine, Jiujiang
  - Jiujiang Third People's Hospital, Jiujiang
  - Jixi Infectious Disease Hospital, Jixi
  - Ji'an Central People's Hospital, Ji’an
  - Karamay Central Hospital, Karamay
  - Yunnan Provincial People's Hospital, Kunming
  - Laixi People's Hospital, Laixi
  - Laizhou People's Hospital, Laizhou
  - Lanzhou Petrochemical General Hospital, Lanzhou
  - Lanzhou Second People's Hospital, Lanzhou
  - The Second Hospital of Lanzhou University, Lanzhou
  - Dongfang Hospital of Lianyungang, Lianyungang
  - Guanyun County Hospital of Traditional Chinese Medicine, Lianyungang
  - Guanyun County People's Hospital, Lianyungang
  - Lianyungang Dongfang Hospital, Lianyungang
  - Lianyungang First People's Hospital, Lianyungang
  - Houma People's Hospital, Linfen
  - Linfen Central Hospital, Linfen
  - Linfen Second People's Hospital, Linfen
  - Linfen Third People's Hospital, Linfen
  - Xiangfen County People's Hospital, Linfen
  - Yaodu District People's Hospital, Linfen
  - Linkou County People's Hospital, Linkou
  - Hezheng County People's Hospital, Linxia
  - Linyi Hospital of Traditional Chinese Medicine, Linyi
  - Linyi People's Hospital, Linyi
  - Lishui Central Hospital, Lishui
  - Liuzhou People's Hospital, Liuchow
  - Liuzhou Workers' Hospital, Liuchow
  - Longnan First People's Hospital, Longnan
  - Liancheng County Hospital, Longyan
  - Longyan People's Hospital, Longyan
  - Longyan Second Hospital, Longyan
  - Tingzhou Hospital of Changting County, Longyan
  - Wuping County Hospital, Longyan
  - Affiliated Hospital of West Anhui Health Vocational College, Lu'an
  - Huoqiu First People's Hospital, Lu'an
  - Huoqiu Second People's Hospital, Lu'an
  - Huoshan County Hospital, Lu'an
  - Jinzhai County Hospital of Traditional Chinese Medicine, Lu'an
  - Lu'an Fourth People's Hospital, Lu'an
  - Lu'an Hospital of Traditional Chinese Medicine, Lu'an
  - Lu'an People's Hospital, Lu'an
  - Lu'an Yeji District People's Hospital, Lu'an
  - Lvliang People's Hospital, Lüliang
  - Wenshui County People's Hospital, Lüliang
  - Macheng People's Hospital, Macheng
  - Huazhou People's Hospital, Maoming
  - Ma'anshan Fourth People's Hospital, Ma’anshan
  - The Second Affiliated Hospital of Wannan Medical College, Ma’anshan
  - Meishan People's Hospital, Meishan
  - Mudanjiang Kang'an Hospital, Mudanjiang
  - Mudanjiang Second People's Hospital, Mudanjiang
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanchang County People's Hospital, Nanchang
  - Nanchang Ninth Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanbu County People's Hospital, Nanchong
  - Nangong People's Hospital, Nangong
  - Jiangsu Provincial People's Hospital, Nanjing
  - Lishui District People's Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Nanjing Hospital of Traditional Chinese Medicine, Nanjing
  - Nanjing Second Hospital, Nanjing
  - Nanjing Tianyinshan Hospital, Nanjing
  - Qinhuai Medical District of Eastern Theater General Hospital, Nanjing
  - The Fourth Affiliated Hospital of Nanjing Medical University, Nanjing
  - Zhongda Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning
  - The Second People's Hospital of Nanning, Nanning
  - Jianyang First Hospital of Nanping, Nanping
  - Nanping First Hospital, Nanping
  - Zhenghe County Hospital, Nanping
  - Affiliated Hospital of Nantong University, Nantong
  - Haimen District People's Hospital, Nantong
  - Nantong Third People's Hospital, Nantong
  - Qidong Third People's Hospital, Nantong
  - Bairin Left Banner People's Hospital, Neimeng
  - Hulunbuir People's Hospital, Neimeng
  - Morin Dawa Daur Autonomous Banner People's Hospital, Neimeng
  - Beilun District Hospital of Traditional Chinese Medicine, Ningbo
  - Ningbo Second Hospital, Ningbo
  - Ningcheng County Central Hospital, Ningcheng
  - Ordos Second People's Hospital, Ordos
  - Panjin Third People's Hospital, Panjin
  - Affiliated Hospital of Gansu Medical College, Pingliang
  - Huating Second People's Hospital, Pingliang
  - Zhuanglang County People's Hospital, Pingliang
  - Pingxiang People's Hospital, Pingxiang
  - Pingyang County People's Hospital, Pingyang
  - Affiliated Hospital of Putian University, Putian
  - Putian First People's Hospital, Putian
  - Putian Hanjiang Hospital, Putian
  - Huangdao District People's Hospital, Qingdao
  - Qingdao Eighth People's Hospital, Qingdao
  - Qingdao Public Health Clinical Center, Qingdao
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Lianzhou People's Hospital, Qingyuan
  - Qingyuan People's Hospital, Qingyuan
  - The Second People's Hospital of Northern Guangdong, Qingyuan
  - Yangshan County People's Hospital, Qingyuan
  - Yingde People's Hospital, Qingyuan
  - Qingzhou People's Hospital, Qingzhou
  - Weifang Yidu Central Hospital, Qingzhou
  - Qinhuangdao Third Hospital, Qinhuangdao
  - The First People's Hospital of Qinzhou, Qinzhou
  - The Second People's Hospital of Qinzhou, Qinzhou
  - Qiqihar Seventh Hospital, Qiqihar
  - Anxi County Hospital of Traditional Chinese Medicine, Quanzhou
  - Anxi County Hospital, Quanzhou
  - Dehua County Hospital of Traditional Chinese Medicine, Quanzhou
  - Huian County Hospital of Traditional Chinese Medicine, Quanzhou
  - Jinjiang Hospital, Quanzhou
  - Nan'an Haidu Hospital, Quanzhou
  - Quangang District Hospital, Quanzhou, Quanzhou
  - Quanzhou Hospital of Traditional Chinese Medicine, Quanzhou
  - Shishi Hospital, Quanzhou
  - The 910th Hospital of the Joint Logistics Support Force, Quanzhou
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou
  - Yongchun County Hospital, Quanzhou
  - Rizhao Central Hospital, Rizhao
  - Rizhao People's Hospital, Rizhao
  - Rui'an Second People's Hospital, Rui’an
  - Ninghua County General Hospital, Sanming
  - Sanming First People's Hospital, Sanming
  - Sanming Hospital of Integrated Traditional Chinese and Western Medicine, Sanming
  - Sanming Second People's Hospital, Sanming
  - Youxi County General Hospital, Sanming, Sanming
  - Youxi County Hospital of Traditional Chinese Medicine, Sanming, Sanming
  - Qilu Hospital of Shandong University, Shandong
  - Shucheng People's Hospital, Shangcheng
  - Minhang District Central Hospital of Shanghai, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai
  - Tongji Hospital Affiliated to Tongji University, Shanghai
  - Shangli County People's Hospital, Shangli
  - Guangxin District People's Hospital, Shangrao
  - Shangrao Central Hospital, Shangrao
  - Shangrao People's Hospital, Shangrao
  - Shangrao Second People's Hospital, Shangrao
  - Wuyuan County People's Hospital, Shangrao
  - Shawan City People's Hospital, Shawan
  - Shengjing Hospital of China Medical University, Shenyang
  - The 242 Hospital Affiliated to Shenyang Medical College, Shenyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Bao'an District People's Hospital, Shenzhen, Shenzhen
  - Bao'an District Traditional Chinese Medicine Hospital, Shenzhen, Shenzhen
  - Fuyong People's Hospital, Bao'an District, Shenzhen, Shenzhen
  - Longgang Central Hospital, Shenzhen, Shenzhen
  - Longgang District People's Hospital, Shenzhen, Shenzhen
  - Longhua District People's Hospital, Shenzhen, Shenzhen
  - Nanshan District People's Hospital, Shenzhen, Shenzhen
  - Peking University Shenzhen Hospital, Shenzhen
  - Shenzhen Fourth People's Hospital, Shenzhen
  - Shenzhen Hospital of Southern Medical University, Shenzhen
  - Shenzhen People's Hospital, Shenzhen
  - Shenzhen Third People's Hospital, Shenzhen
  - Songgang People's Hospital, Bao'an District, Shenzhen, Shenzhen
  - Southern Medical University Shenzhen Hospital, Shenzhen
  - The Eighth Affiliated Hospital of Sun Yat-sen University, Shenzhen
  - The Seventh Affiliated Hospital of Sun Yat-sen University, Shenzhen
  - Yantian District People's Hospital, Shenzhen, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Sinopharm Dongfeng General Hospital, Shiyan
  - Shouguang People's Hospital, Shouguang
  - Qionglai Medical Center Hospital, Sichuan
  - Songyuan Jilin Oilfield Hospital, Songyuan
  - Nanjing Drum Tower Hospital Group, Suqian
  - Shuyang County Hospital of Traditional Chinese Medicine, Suqian
  - Sihong First People's Hospital, Suqian
  - Suqian First People's Hospital, Suqian
  - Suqian Hospital Affiliated to Nanjing Drum Tower Hospital Group, Suqian
  - Suqian Zhongwu Hospital, Suqian
  - he First Affiliated Hospital of Soochow University, Suzhou
  - Kunshan First People's Hospital, Suzhou
  - Kunshan Hospital of Traditional Chinese Medicine, Suzhou
  - Rudong County People's Hospital, Suzhou
  - Suzhou Fifth People's Hospital, Suzhou
  - Suzhou Hospital of Integrated Traditional Chinese and Western Medicine, Suzhou
  - Suzhou Municipal Hospital, Suzhou
  - Suzhou Ninth People's Hospital, Suzhou
  - Taicang First People's Hospital, Suzhou
  - The Fourth Affiliated Hospital of Soochow University, Suzhou
  - Xiaoxian People's Hospital, Suzhou
  - Zhangjiagang First People's Hospital, Suzhou
  - Taihe County People's Hospital, Taihe
  - Shanxi Bethune Hospital, Taiyuan
  - Shanxi Provincial Hospital of Traditional Chinese Medicine, Taiyuan
  - Shanxi Provincial People's Hospital, Taiyuan
  - Taiyuan Central Hospital, Taiyuan
  - Taiyuan Third People's Hospital, Taiyuan
  - The First Hospital of Shanxi Medical University, Taiyuan
  - Taixing People's Hospital, Taizhou
  - Taixing Second People's Hospital, Taizhou
  - Taizhou People's Hospital, Taizhou
  - Taizhou Second People's Hospital, Taizhou
  - Xinghua People's Hospital, Taizhou
  - Zhejiang Taizhou Hospital, Taizhou
  - Tai'an Central Hospital, Tai’an
  - Tangshan Seventh Hospital, Tangshan
  - Tengzhou Central People's Hospital, Tengzhou
  - Baodi District People's Hospital, Tianjin
  - Binhai New Area Dagang Hospital, Tianjin
  - Tianjin Binhai People's Hospital, Tianjin
  - Tianjin Fifth Central Hospital, Tianjin
  - Tianjin Port Hospital, Tianjin
  - Tianjin Second People's Hospital, Tianjin
  - Tianjin TEDA Hospital, Tianjin
  - Tianjin Third Central Hospital, Tianjin
  - Tongjiang People's Hospital, Tongjiang
  - Tongliao Sixth People's Hospital, Tongliao
  - Tongling People's Hospital, Tongling
  - The Fifth Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Xinjiang Uyghur Autonomous Region Traditional Chinese Medicine Hospital, Ürümqi
  - Weifang People's Hospital, Weifang
  - The 970th Hospital of the Joint Logistics Support Force, PLA, Weihai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wenzhou Sixth People's Hospital, Wenzhou
  - Wuhai Fifth People's Hospital, Wuhai
  - Changjiang Shipping General Hospital (Wuhan Brain Hospital), Wuhan
  - Hubei Third People's Hospital (Hubei Zhongshan Hospital), Wuhan
  - Jiangxia District First People's Hospital, Wuhan, Wuhan
  - The Fifth Hospital of Wuhan, Wuhan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuhan Hankou Hospital, Wuhan
  - Wuhan Jinyintan Hospital, Wuhan
  - Wuhan Seventh Hospital, Wuhan
  - Gansu Wuwei Cancer Hospita, Wuwei
  - Wuwei People's Hospital, Wuwei
  - Jiangyin People's Hospital, Wuxi
  - Jiangyin Traditional Chinese Medicine Hepatobiliary Hospital, Wuxi
  - Taihu Hospital, Wuxi
  - Wuxi Fifth People's Hospital, Wuxi
  - Wuxi No. 2 Hospital of Traditional Chinese Medicine, Wuxi
  - Wuxi No. 5 People's Hospital, Wuxi
  - Wuxi Second Hospital of Traditional Chinese Medicine, Wuxi
  - Yixing People's Hospital, Wuxi
  - The Third People's Hospital of Wuzhou, Wuzhou
  - Wu'an First People's Hospital, Wu’an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The 909th Hospital of the Joint Logistics Support Force, Xiamen
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen
  - Zhongshan Hospital Xiamen, Fudan University, Xiamen
  - Xiaogan Central Hospital, Xiaogan
  - Yunmeng County People's Hospital, Xiaogan
  - Qinghe County People's Hospital, Xingtai
  - Xingtai Fifth Hospital, Xingtai
  - Xingtai Ninth Hospital, Xingtai
  - Xingtai People's Hospital, Xingtai
  - Datong Hui and Tu Autonomous County People's Hospital, Xining
  - Qinghai Fourth People's Hospital, Xining
  - Qinghai Provincial People's Hospital, Xining
  - Qinghai Red Cross Hospital, Xining
  - Ili Kazakh Autonomous Prefecture Kuitun Hospital, Xinjiang
  - Xinjiang Production and Construction Corps 6th Division Hospital, Xinjiang
  - Xintai People's Hospital, Xintai
  - Xiushui County First People's Hospital, Xiushui
  - People's Hospital of Tibet Autonomous Region, Xizang
  - Shannan People's Hospital, Xizang
  - Third People's Hospital of Tibet Autonomous Region, Xizang
  - Jixi County People's Hospital, Xuancheng
  - Xuancheng Central Hospital, Xuancheng
  - Xuancheng People's Hospital, Xuancheng
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Feng County People's Hospital, Xuzhou
  - Pei County People's Hospital, Xuzhou
  - Pizhou People's Hospital, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Xuzhou Infectious Disease Hospital, Xuzhou
  - Xuzhou Mining Group Traditional Chinese Medicine Hospital, Xuzhou
  - Xuzhou New Health Hospital, Xuzhou
  - Yan'an Hospital of Traditional Chinese Medicine, Yanan
  - Yan'an People's Hospital, Yanan
  - Affiliated Hospital of Yanbian University, Yanbian
  - Dunhua City Hospital, Yanbian
  - Wangqing County People's Hospital, Yanbian
  - Funing County People's Hospital, Yancheng
  - Jianhu County People's Hospital, Yancheng
  - Xuyi County People's Hospital, Yancheng
  - Yancheng First People's Hospital, Yancheng
  - Yancheng Seventh People's Hospital, Yancheng
  - Yangquan Coal Mining Group General Hospital, Yangquan
  - Yangquan Third People's Hospital, Yangquan
  - Jiangdu District Third People's Hospital, Yangzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yangzhou Third People's Hospital, Yangzhou
  - Binzhou Medical University Yantai Affiliated Hospital, Yantai
  - Yantai Qishan Hospital, Yantai
  - Yibin First People's Hospital, Yibin
  - Dangyang People's Hospital, Yichang
  - Yichang Central People's Hospital, Yichang
  - Yichang Third People's Hospital, Yichang
  - Zhijiang People's Hospital, Yichang
  - Yichun People's Hospital, Yichun
  - Ningxia Medical University General Hospital, Yinchuan
  - Yingkou Third People's Hospital, Yingkou
  - Yingtan People's Hospital, Yingtan
  - Ili Kazakh Autonomous Prefecture Traditional Chinese Medicine, Yining
  - Yining City People's Hospital, Yining
  - Jingbian County People's Hospital, Yulin
  - The First People's Hospital of Yulin, Yulin
  - The Second People's Hospital of Yulin, Yulin
  - Yulin First Hospital, Yulin
  - Yulin Hospital of Traditional Chinese Medicine, Yulin
  - Jishan County People's Hospital, Yuncheng
  - Linyi County People's Hospital, Yuncheng
  - Xia County People's Hospital, Yuncheng
  - Yanhu District People's Hospital, Yuncheng City, Yuncheng
  - Yongji People's Hospital, Yuncheng
  - Yuncheng Hospital of Traditional Chinese Medicine, Yuncheng
  - Yuncheng Second Hospital, Yuncheng
  - Shandong Health Group Zaozhuang Central Hospital, Zaozhuang
  - Zhangjiakou Infectious Disease Hospital, Zhangjiakou
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
  - Jurong People's Hospital, Zhenjiang
  - Yangzhong Hospital of Traditional Chinese Medicine, Zhenjiang
  - Yangzhong People's Hospital, Zhenjiang
  - Zhenjiang Third People's Hospital, Zhenjiang
  - The Second People's Hospital of Zhongshan, Zhongshan
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan
  - Zibo City No.148 Hospital, Zibo
  - Zibo Hospital of Traditional Chinese Medicine, Zibo
  - Zibo Infectious Diseases Hospital, Zibo
  - Zigong First People's Hospital, Zigong